CLINICAL TRIAL: NCT02753608
Title: Exhalate Sample Collection for Raman Spectroscopy-based Early Detection of Ventilator-associated Pneumonia (VAP)
Brief Title: Early Detection of Ventilator-associated Pneumonia (VAP)
Acronym: cheqVAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jena University Hospital (Other)
Responsible Party: Principal Investigator, Mathias Pletz, Director, Center for Infection Medicine and Hospital Hygiene, Jena University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ZKSJ0093
Record Dates: First submitted 2016-03-31; First posted 2016-04-28 (Estimated); Last update posted 2018-07-20 (Actual); Status verified 2018-07

CONDITIONS: Pneumonia, Ventilator-associated
Keywords: exhaled breath condensate; volatile organic compounds
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- No ventilator-associated pneumonia (VAP) (Sham Comparator): Collection of exhaled breath condensate (EBC) in patients without clinical signs of VAP
  Interventions: Other: Collection of exhaled breath condensate
- Ventilator-associated pneumonia (VAP) (Experimental): Collection of exhaled breath condensate (EBC) in patients displaying clinical signs of VAP
  Interventions: Other: Collection of exhaled breath condensate

INTERVENTIONS:
Other: Collection of exhaled breath condensate — An sampling device (authorized for this use) will be connected to the expiratory line of the ventilator. Exhaled breath condensates accumulate in a cooled container.
  Other Names: EBC collection

SUMMARY:
The study goal consists in the sequential collection of exhaled breath condensates (EBC) from patients receiving invasive ventilation. Subsequent Raman spectroscopy aims at the identification of putative biomarkers that could enable rapid early distinction of Ventilator-associated pneumonia.

DETAILED DESCRIPTION:
Diagnostics of VAP relies on two complementary strategies: meeting pre-defined clinical criteria and evidence of pathogens in the lower respiratory tract. Mere reliance on clinical symptoms, such as radiologic evidence, systemic signs of inflammation and indices of compromised pulmonary function reportedly lead to misdiagnosis. Current diagnostic procedures recommend gathering of evidence for new or progressive lung infiltrates from serial chest radiographies, together with co-existing clinical signs of impaired respiratory function. Microbiological confirmation of pathogen presence requires examination of airway secretions collected by invasive bronchoalveolar lavage which demands specific technical skills and staff training. Although verification of causal pathogens is essential for the introduction of targeted antibiotic therapy, the procedure is time-consuming and qualitative in reportedly less than 30 % of the cases. Furthermore, the currently adopted diagnostic approaches are based on sporadic information sampling and do not support continuous monitoring and evaluation of the effect of therapeutic interventions. All above-listed flaws and shortcomings emphasize the need for rapid, reliable and non-invasive recognition of VAP, preferably in a setting that would permit continuous bedside monitoring and timely introduction of targeted drug therapy.

The study objective consists in sequential collection of exhaled breath condensates (EBC) in ICU patients receiving invasive ventilation. The EBC samples will be subjected to determination of volatile organic compound (VOC) profiles by Stimulated Raman Spectroscopy (SRS) which, upon individual matching to routinely collected clinical parameters, may become putative biomarkers for the early recognition of VAP. Evidence has accumulated in support of the assumption that certain metabolites in EBC might display significant profile differences as to their size, hydrophobicity and electrical charge. Identification of VAP-specific profiles of VOC will provide the basis for the generation of a data base enabling the construction and standardization of a bedside device for continuous real-time point-of-care monitoring of VAP hazard in patients on invasive ventilation.

ELIGIBILITY:
Inclusion Criteria:

* ICU patients on invasive ventilation
* Signed informed consent

Exclusion Criteria:

* Glucocorticoid dosage above 0.3 mg/kg Prednisolone equivalent over more than 3 weeks
* Treatment with recognized T cell immunosuppressant (cyclosporine, Tumor Necrosis Factor antagonists) or nucleoside analogues during the preceding 90 days
* Inherited severe immunodeficiency
* Solid organ or stem cell transplant recipients
* Anti-cancer chemotherapy during the preceding 90 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-06-28 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Raman spectra of volatile organic compounds in exhaled breath condensates in the absence or presence of VAP | 24 hours upon clinical diagnosis confirmation
  Raman spectrum of volatile organic compounds

CONTACTS AND LOCATIONS:
Overall Officials: Mathias Pletz, MD, Principal Investigator — Jena University Hospital
Locations (1):
- Jena University Hospital, Jena, Thuringia, Germany

IPD SHARING:
Plan to Share IPD: No
Individual participant data will be not made available